CLINICAL TRIAL: NCT03253601
Title: iADAPT to Support Strategy Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Elizabeth R. Skidmore, PhD, OTR/L, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO17030372
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Adherence, Patient; Strategy Training
Keywords: Rehabilitation; Disability; Mobile Health Technology
MeSH Terms: conditions — Stroke; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy Training: iADAPT Application (Experimental): Participants will use the iADAPT mobile health application to supplement to in-person and remote intervention sessions.
  Interventions: Behavioral: Strategy Training
- Strategy Training: Workbook (Active Comparator): Participants will use a printed workbook to supplement to in-person and remote (by telephone) intervention sessions.
  Interventions: Behavioral: Strategy Training

INTERVENTIONS:
Behavioral: Strategy Training — Strategy training is a form of meta-cognitive instruction that trains individuals with stroke-related cognitive impairments to identify and prioritize problematic daily activities, identify the barriers impeding performance, generate and evaluate their own strategies to address barriers, and apply these skills through iterative practice.

SUMMARY:
Adherence to rehabilitation interventions is associated with functional outcomes (e.g. independence in daily activities, return of motor function) after stroke. Low adherence to rehabilitation home programs is common after stroke. Interventions delivered via mobile health applications demonstrated positive effects on adherence to health behaviors (e.g. medication routines, smoking cessation). The investigators developed the iADAPT mobile application to support adherence to Strategy Training. Strategy Training is an iterative rehabilitation intervention the promotes goal setting, planning, and self-monitoring after stroke. This study examines the effects of the iADAPT mobile health application relative to a workbook on adherence to Strategy Training after stroke.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of Stroke

Exclusion Criteria:

* prior exposure to Strategy Training
* vision impairment that impairs ability to read device screen or worksheet
* poor self-awareness (score of ≥2 on Self Awareness of Deficits Inventory item #1 or #2
* current major depressive, bipolar, or psychotic disorder (Patient Health Questionnaire-9, PRIME-MD)
* current alcohol or drug abuse (Mini International Neuropsychiatric Interview)
* severe aphasia (score ≤1 on Boston Diagnostic Aphasia Examination)
* current diagnosis of dementia, neurodegenerative disease, or cancer
* anticipated discharge to a skilled nursing facility

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence: Observed client behavior | Baseline to 3 months
  Number of completed activity trials in the iADAPT application or Workbook
Adherence: Client-reported progress on goals. | Baseline and 3 months
  Client rating of independence with self-selected goals (measured using Canadian Occupational Performance Measure)

SECONDARY OUTCOMES:
Adherence: Client perspectives on treatment environment | Baseline and 3 months
  Client rating on patient-provider connection and treatment expectancy measured by Healing Encounters and Attitudes Lists

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R. Skidmore, PhD, OTR/L, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No